CLINICAL TRIAL: NCT02360462
Title: The Effect of tDCS in the Preoperative Period of Hallux Valgus Surgical Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Hospital Independencia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-0643
Record Dates: First submitted 2015-01-22; First posted 2015-02-10 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Chronic Pain; Hallux Valgus
Keywords: Transcranial Direct Current Stimulation; tDCS; Hallux Valgus; Chronic Pain
MeSH Terms: conditions — Chronic Pain; Hallux Valgus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): Active tDCS will be applied in the head of the patients in 20 minute sessions, twice. First session will be applied in the night before and the second session, in the morning before the surgical procedure. The stimulation will be administered with a pair of surface electrodes, sponge coated, soaked in saline. A battery-powered constant current stimulator will be used for this purpose (tDCS device). The stimulation is performed by placing the anodal electrode in the primary motor cortex (M1) and the cathodal one in the contralateral supraorbital area, and it will use a 2 mA current
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): The sham tDCS consists in the same montage of the active tDCS, but the device is turned off 30 seconds after starting stimulation (without letting the patient notice it). The rest of the montage is kept identical to the active one during the 20 minutes session.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — The stimulation will be administered with a pair of surface electrodes, sponge coated, soaked in saline. A battery-powered constant current stimulator will be used for this purpose (tDCS device). The stimulation is performed by placing the anodal electrode in the primary motor cortex (M1) and the cathodal one in the contralateral supraorbital area and it will use a 2 mA (milliampere) current.
  Other Names: transcranial direct current stimulation (tDCS)
  Arms: Active tDCS
Device: Sham tDCS — The sham tDCS consists in the same montage of the active tDCS, but the device is turned off 30 seconds after stimulation starts (without letting the patient notice it). The rest of the montage is kept identical to the active one during the 20 minutes session
  Other Names: Sham transcranial direct current stimulation (Sham tDCS)
  Arms: Sham tDCS

SUMMARY:
This is a clinical trial that intend to determine if transcranial direct current stimulation (tDCS) is effective in the treatment of postoperative pain and in the anxiety level in the preoperative period of hallux valgus surgical treatment

DETAILED DESCRIPTION:
Introduction: Forefoot deformities are important cause of feet pain and discomfort and affect around 80% of general population, predominantly in female population. Among teenagers and adults´ common forefoot deformities is hallux valgus. To achieve the deformity heal, surgical treatment is needed. The transcranial direct current stimulation (tDCS) is a non invasive technic, that aims for the central nervous system modulation for pain control, which can become a therapeutic option for postoperative pain. Experimental studies have shown that tDCS has reverted the hyperalgesia induced by chronic stress and articular inflammatory pain, has reduced total knee arthroplasty postoperative opioid consumption and a single 20 minutes session has shown reduction in endoscopic procedures opioid consumption, safety and minimal adverse effects. However, the tDCS effect in preoperative hyperalgesia has not been explored yet in sensitized patients, neither in anxiety and postoperative rehabilitation of patients submitted to hallux valgus surgical correction. In this study, it was chosen to use tDCS to stimulate cerebral cortex due to its efficacy in painful syndromes, for being a non invasive, low cost and easy-to-apply technic in comparison to other neurostimulation technics and especially, for its potential to counter-regulate the mal adaptive neuroplastic alterations associated to chronic pain. Objective: to evaluate the effect of tDCS compared to tDCS-sham in the pain control (visual analog scale score, pain threshold and the descendent modulator system), perioperative anxiety, postoperative analgesic drug consumption and in the rehabilitation of patients with arthralgia of the first metatarsophalangeal articulation submitted to hallux valgus surgical correction. Method: it is a randomized, blinded, placebo-sham controlled clinical trial which includes 40 female patients, between 18 and 70 years old, candidates to hallux valgus surgical treatment by combined Chevron + Akin osteotomy due to arthralgia of the first metatarsophalangeal articulation. The patients will be randomized and divided into two groups that will be treated with two tDCS or tDCS-sham sessions of 20 minutes each in preoperative period. Expected results: This study will evaluate the effect of tDCS as a treatment option to postoperative pain and perioperative anxiety of patients submitted to hallux valgus surgical correction. In case of proven efficacy, this technic can become a low cost, easy access, safe and effective treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

* indication of hallux valgus surgical treatment because of arthralgia of the first metatarsophalangeal joint,
* capability of writing and understanding the Portuguese language

Exclusion Criteria:

* diabetic neuropathy,
* history of intense or frequent headache,
* chronic dermatologic disease,
* previous adverse effects to treatment with tDCS, seizures,
* severe cranial trauma with alteration of the cranial anatomy,
* metallic intracranial implants or pacemaker,
* non-compensated psychiatric disease,
* non-collaborative patients,
* history of neurologic,
* oncologic disease,
* heart, renal or hepatic failure.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in pain scores assessed with the visual analogue scale | Once Daily. It starts in the day before surgical treatment (Day 0), and it is assessed every day until one week after the surgical procedure (total = 10 days)
  Patients will be asked their worst pain level (assessed by the Visual Analogue Scale) with 2 different scores: worst daily pain including movement period and pain in rest period. It will also be assessed a pain score for the moment before and another for the moment right after each tDCS session (Day 0 and Day 1). The outcome assessor will visit the patient once daily during the hospital stay (an expected average of 2 days) and will call the patient once daily after discharge. Patients will also be asked to daily write down the analgesic drug intake after hospital discharge and the outcome assessor will review nursery notes during hospital stay for drug intake. Total evaluations: 10 days

SECONDARY OUTCOMES:
Preoperative Anxiety level | Initial contact (before any tDCS session - Day 0) and the moment before the surgical procedure (Day 1)
  Anxiety level will be assessed by State-Trait Anxiety Inventory (STAI), adapted to Brazilian Portuguese Language. It will be assessed before the first session of tDCS (on initial contact with the patient - Day 0), and in the moment right before going to the surgical room in the next day (Day 1). Total = 2 evaluations
Change in the temperature pain threshold | Day before the surgical treatment (Day 0), and in the moment after the spinal anesthesia recovery in immediate postoperative period (Day 1).
  It will be assessed by the Quantitative Sensory Test (QST) in the dominant (right) forearm and in the leg ipsilateral to the foot that will be treated. The heat pain tolerance, the pain threshold to the heat and the temperature defined as pain 6/10 by the participant will be determined. The temperature starts at 32°C, and it heats at a 1.0 °C/sec rate and cools down after a button is pressed or whenever it reaches the max temperature of 52°C. The participant will be asked to press down the button at the first sensation of pain to determine the pain threshold; to press down the button whenever she can not stand the heat anymore for the pain tolerance determination and, for last, to press down the button at the temperature she fells pain equivalent to 6/10 in the numeric scale of pain. The pain threshold and the temperature of pain 6/10 will be determined by the arithmetic mean of 3 evaluations each.
Change in effect of the descendent modulator system of pain | Day before the surgical treatment (Day 0), and in the moment after the spinal anesthesia recovery in immediate postoperative period (Day 1).
  It will be assessed by the Conditioned Pain Modulation test (CPM). A nociceptive tonic conditioning stimulus - immersion of the non-dominant hand in cold water (0°C for 1 minute) - will be applied concomitant to the progressive thermal stimulus in the dominant forearm as applied in the QST pattern until it reaches the 6/10 pain temperature previously determined by the participant. It will be tested in the day before the surgical treatment (before the first session of tDCS), and after the spinal anesthesia recovery in immediate postoperative period. Total of 2 test days.
Change in serum biomarkers level: The brain derived neurotrophic factor (BDNF), S100B, nerve growth factor (NGF) and enolase | The day before the surgical treatment (Day 0), in the moment before the spinal anestesia (Day 1) and a week after the surgical procedure (Day 9)
  A blood sample will be collected to measure each plasma biomarker in the day before the surgical treatment (Day 0), in the moment before the spinal anesthesia (Day 1) and a week after the surgical procedure (Day 9). Total = 3 evaluations

OTHER OUTCOMES:
Adverse Effects | At the end of each tDCS session (Day 0 and Day 1)
  At the end of each tDCS session, the incidence of any adverse effects - paresthesia, headache, dizziness, nausea, neck pain, burns, redness or pain in the scalp, insomnia, abrupt humor changes and lack of concentration - will be questioned to the participant. Total = 2 evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital Independência, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valle A, Roizenblatt S, Botte S, Zaghi S, Riberto M, Tufik S, Boggio PS, Fregni F. Efficacy of anodal transcranial direct current stimulation (tDCS) for the treatment of fibromyalgia: results of a randomized, sham-controlled longitudinal clinical trial. J Pain Manag. 2009;2(3):353-361. PMID 21170277
- [Background] Boros K, Poreisz C, Munchau A, Paulus W, Nitsche MA. Premotor transcranial direct current stimulation (tDCS) affects primary motor excitability in humans. Eur J Neurosci. 2008 Mar;27(5):1292-300. doi: 10.1111/j.1460-9568.2008.06090.x. Epub 2008 Feb 29. PMID 18312584
- [Background] Nitsche MA, Liebetanz D, Antal A, Lang N, Tergau F, Paulus W. Modulation of cortical excitability by weak direct current stimulation--technical, safety and functional aspects. Suppl Clin Neurophysiol. 2003;56:255-76. doi: 10.1016/s1567-424x(09)70230-2. No abstract available. PMID 14677403
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Fenton BW, Palmieri PA, Boggio P, Fanning J, Fregni F. A preliminary study of transcranial direct current stimulation for the treatment of refractory chronic pelvic pain. Brain Stimul. 2009 Apr;2(2):103-7. doi: 10.1016/j.brs.2008.09.009. Epub 2009 Feb 28. PMID 20633407
- [Background] Caumo W, Ruehlman LS, Karoly P, Sehn F, Vidor LP, Dall-Agnol L, Chassot M, Torres IL. Cross-cultural adaptation and validation of the profile of chronic pain: screen for a Brazilian population. Pain Med. 2013 Jan;14(1):52-61. doi: 10.1111/j.1526-4637.2012.01528.x. Epub 2012 Nov 21. PMID 23171145
- [Background] Sehn F, Chachamovich E, Vidor LP, Dall-Agnol L, de Souza IC, Torres IL, Fregni F, Caumo W. Cross-cultural adaptation and validation of the Brazilian Portuguese version of the pain catastrophizing scale. Pain Med. 2012 Nov;13(11):1425-35. doi: 10.1111/j.1526-4637.2012.01492.x. Epub 2012 Oct 4. PMID 23036076
- [Derived] Ribeiro H, Sesterhenn RB, Souza A, Souza AC, Alves M, Machado JC, Burger NB, Torres ILDS, Stefani LC, Fregni F, Caumo W. Preoperative transcranial direct current stimulation: Exploration of a novel strategy to enhance neuroplasticity before surgery to control postoperative pain. A randomized sham-controlled study. PLoS One. 2017 Nov 30;12(11):e0187013. doi: 10.1371/journal.pone.0187013. eCollection 2017. PMID 29190741